CLINICAL TRIAL: NCT04826354
Title: Effects of High-dose StAtin Versus Low-dose Statin Plus Ezetimibe on Statin-Associated Muscle Symptoms & on Reaching Target LDL-C Levels Among Elderly Patients With Atherosclerotic Cardiovascular Disease
Brief Title: Effects of Statin for Elderly Patients With Atherosclerotic Cardiovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaveSAMS
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Atheroscleroses, Coronary
Keywords: Elderly; Statin; Ezetimibe
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Effects of high-dose Statin Versus low-dose statin plus ezetimibe on statin-associated Muscle Symptoms
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin
- Rosuvamibe (Active Comparator): Rosuvastatin plus ezetimibe 10/5
  Interventions: Drug: Rosuvastatin and Ezetimibe

INTERVENTIONS:
Drug: Rosuvastatin and Ezetimibe — Rosuvastatin Versus Rosuvastatin plus Ezetimibe
  Arms: Rosuvamibe
Drug: Rosuvastatin — Rosuvastatin
  Arms: Rosuvastatin

SUMMARY:
High-dose statins can reduce mortality and cardiovascular events in patients with established atherosclerotic cardiovascular disease (ASCVD). Therefore, US and European recommendations recommend that established ASCVD patients (coronary artery disease, cerebrovascular disease, peripheral vascular disease) use high-dose statins to lower LDL cholesterol levels by at least 50%. However, in actual practice, high-dose statins are relatively less used, and the reason is unclear, but it is believed to be due to concerns about the side effects of high-dose statins. Most of the side effects of statins are statin-associated muscle symptoms (SAMS), which are more common than the incidence in clinical studies, especially in frontline care. These muscle side effects are dose-dependent and are common at high doses, and the incidence is known to increase in the elderly over 70 years of age. However, the US recommendation recommends using high-dose statins to lower LDL cholesterol by 50% or more to prevent cardiovascular events even in ASCVD patients over 70 years of age.

Most early studies on lowering LDL cholesterol in ASCVD patients used high doses of statins. However, after introducing cholesterol absorption inhibitors ezetimibe and PCSK9 inhibitor, large-scale clinical studies have been conducted to lower LDL cholesterol using these drugs. In this study, as in the statin study, cardiovascular events were significantly reduced, and together with statins, it became a standard treatment for ASCVD patients. On the other hand, the clinical benefit shown in clinical studies using cholesterol-lowering agents so far depends entirely on how much LDL cholesterol is lowered and how long it is maintained in a low state, indicating that LDL cholesterol management is the core of arteriosclerosis treatment. In addition to high-dose statins, a combination of low-dose statins and ezetimibe can be cited as a method for lowering LDL cholesterol to more than 50%. In the latter case, it is expected that there will be an advantage of reducing muscle side effects by reaching the target LDL cholesterol level by using a low-dose statin. However, no studies compare the difference in muscle side effects between low-dose statins and ezetimibe combination drugs, which reduce LDL cholesterol to the same extent compared to high-dose statins, in elderly patients over 70 years of age with ASCVD. In this study, the association of low-dose rosuvastatin 5mg and ezetimibe combination (rosuvastatin 10/5mg) compared to high-dose rosuvastatin 20mg in elderly patients 70 years of age or older with established ASCVD. This study aims to compare and analyze the incidence of muscle symptoms (SAMS) and their effect on LDL cholesterol.

DETAILED DESCRIPTION:
Established Atherosclerotic Cardiovascular Disease (ASCVD)

A. Coronary artery disease meeting at least one of the following criteria:

* A history of coronary recanalization in multivessel coronary artery disease, evidenced by any of the following:

  1. Percutaneous coronary intervention (PCI) of one or more vessels, including branching arteries
  2. PCI or coronary artery bypass grafting (CABG) for >50% residual stenosis in separate vessels that have not undergone recanalization
  3. multivessel CABG at least 5 years prior to screening
* Significant coronary without prior revascularization, evidenced by >70% stenosis in at least one coronary artery, >50% stenosis in two or more coronary arteries, or >50% stenosis in the left main coronary artery arterial disease
* Known coronary calcium score > 100 in subjects who did not undergo coronary recanalization prior to randomization

B. Cerebrovascular Disease meeting at least one of the following criteria:

* Previous transient ischemic attack with carotid artery stenosis in 50%
* 70% internal or external carotid artery stenosis or >50% stenosis of two or more
* Past history of recanalization of internal or external carotid artery

C. Peripheral arterial disease meeting at least one of the following criteria:

* > 50% stenosis in the arteries of the extremities
* History of abdominal aortic treatment (percutaneous or surgical) for atherosclerotic disease
* Ankle Brachial Index (ABI) ≤ 0.90

ELIGIBILITY:
Inclusion Criteria (must satisfy all of the following selection criteria) :

1. Those who are 70 years of age or older as of the date of consent
2. Established arteriosclerotic cardiovascular disease (coronary artery disease, cerebrovascular disease, or peripheral vascular disease)
3. Subjects who have consented to the study plan and follow-up observation by the patient or representative, and who consented in advance in writing to the clinical subject consent approved by the research deliberation committee/ethics committee of the research institution

Exclusion Criteria:

1. Take statins or ezetimibe within the last 4 weeks
2. In case of end-stage kidney disease (eGFR<30 ml/min/1.73m2)
3. Heart surgery or major surgery is planned within the next 6 months
4. Patients with chronic diseases such as severe lung disease, stroke, etc.
5. Patients with chronic inflammatory diseases who require oral, intravenous, or intra-articular steroid treatment (Ointments, inhalants, or intranasal steroids are allowed)
6. If you have been diagnosed with cancer within the past 1 year or are currently receiving chemotherapy
7. In the case of clinically significant abnormal findings that may infringe on the safety of the study by the investigator's judgment confirmed in a screening visit, physical examination, blood test, or electrocardiogram
8. Liver disease, bile duct obstruction, or liver enzyme level (ALT/AST) is more than 3 times normal
9. If you have a disease whose life expectancy is less than 1 year
10. If you do not want or cannot comply with the procedure described in the research proposal

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 582 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Statin-Associated Muscle Symptoms (SAMS) | 6 month
  Patients with a Proposed Statin Myalgia Index score of 7 or higher (Cardiovasc Drugs Ther 2003;17:459-465):
  * Aspects: muscle pain, muscle spasms, muscle stiffness, feeling of strength, ligament pain, etc.
  * Location: thigh, buttocks, calves, back muscle, proximal arms
  * Onset time after dosing: within 6 months
  * Deteriorating factors: exercise, rest, cold exposure, position change, fasting
  * Severe: Occurs in abnormalities in daily life, occurs in daily life, occurs in less than daily life
Target Low density lipoprotein cholesterol (LDL-C) achievement | 6 month
  Target LDL-C achievement (LDL <70mg/dL)

SECONDARY OUTCOMES:
CK levels | 6 month
  Creatinine Kinase levels
GOT levels | 6 month
  Aspartate Transaminase (Glutamic Oxaloacetic Transaminase levels
GPT levels | 6 month
  Alanine Transaminase (Glutamic Pyruvic Transaminase) levels
Levels of Total cholesterol, LDL cholesterol, HDL cholesterol | 6 month
  Levels of Total cholesterol, LDL cholesterol, HDL cholesterol
Level of Triglyceride | 6 month
  Level of Triglyceride
Level of high sensitive-CRP | 6 month
  Level of high sensitive-CRP
Incidence of myopathy, rhabdomyolysis | 6 month
  Incidence of myopathy, rhabdomyolysis
Frequency of drug discontinuation due to SAMS side effects | 6 month
  Frequency of drug discontinuation due to SAMS side effects
Frequency of drug discontinuation due to side effects other than SAMS | 6 month
  Frequency of drug discontinuation due to side effects other than SAMS

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul

REFERENCES:
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Ference BA, Ginsberg HN, Graham I, Ray KK, Packard CJ, Bruckert E, Hegele RA, Krauss RM, Raal FJ, Schunkert H, Watts GF, Boren J, Fazio S, Horton JD, Masana L, Nicholls SJ, Nordestgaard BG, van de Sluis B, Taskinen MR, Tokgozoglu L, Landmesser U, Laufs U, Wiklund O, Stock JK, Chapman MJ, Catapano AL. Low-density lipoproteins cause atherosclerotic cardiovascular disease. 1. Evidence from genetic, epidemiologic, and clinical studies. A consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2017 Aug 21;38(32):2459-2472. doi: 10.1093/eurheartj/ehx144. PMID 28444290
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):3168-3209. doi: 10.1016/j.jacc.2018.11.002. Epub 2018 Nov 10. No abstract available. PMID 30423391
- [Background] European Association for Cardiovascular Prevention & Rehabilitation; Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines (CPG) 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28. PMID 21712404
- [Background] Pokharel Y, Tang F, Jones PG, Nambi V, Bittner VA, Hira RS, Nasir K, Chan PS, Maddox TM, Oetgen WJ, Heidenreich PA, Borden WB, Spertus JA, Petersen LA, Ballantyne CM, Virani SS. Adoption of the 2013 American College of Cardiology/American Heart Association Cholesterol Management Guideline in Cardiology Practices Nationwide. JAMA Cardiol. 2017 Apr 1;2(4):361-369. doi: 10.1001/jamacardio.2016.5922. PMID 28249067
- [Background] Rodriguez F, Lin S, Maron DJ, Knowles JW, Virani SS, Heidenreich PA. Use of high-intensity statins for patients with atherosclerotic cardiovascular disease in the Veterans Affairs Health System: Practice impact of the new cholesterol guidelines. Am Heart J. 2016 Dec;182:97-102. doi: 10.1016/j.ahj.2016.09.007. Epub 2016 Sep 29. PMID 27914506
- [Background] Rosenson RS, Kent ST, Brown TM, Farkouh ME, Levitan EB, Yun H, Sharma P, Safford MM, Kilgore M, Muntner P, Bittner V. Underutilization of high-intensity statin therapy after hospitalization for coronary heart disease. J Am Coll Cardiol. 2015 Jan 27;65(3):270-7. doi: 10.1016/j.jacc.2014.09.088. PMID 25614424
- [Background] Riphagen IJ, van der Veer E, Muskiet FA, DeJongste MJ. Myopathy during statin therapy in the daily practice of an outpatient cardiology clinic: prevalence, predictors and relation with vitamin D. Curr Med Res Opin. 2012 Jul;28(7):1247-52. doi: 10.1185/03007995.2012.702102. Epub 2012 Jun 28. PMID 22686958
- [Background] Bruckert E, Hayem G, Dejager S, Yau C, Begaud B. Mild to moderate muscular symptoms with high-dosage statin therapy in hyperlipidemic patients--the PRIMO study. Cardiovasc Drugs Ther. 2005 Dec;19(6):403-14. doi: 10.1007/s10557-005-5686-z. PMID 16453090
- [Background] Armitage J. The safety of statins in clinical practice. Lancet. 2007 Nov 24;370(9601):1781-90. doi: 10.1016/S0140-6736(07)60716-8. PMID 17559928
- [Background] Nguyen KA, Li L, Lu D, Yazdanparast A, Wang L, Kreutz RP, Whipple EC, Schleyer TK. A comprehensive review and meta-analysis of risk factors for statin-induced myopathy. Eur J Clin Pharmacol. 2018 Sep;74(9):1099-1109. doi: 10.1007/s00228-018-2482-9. Epub 2018 May 22. PMID 29785580
- [Background] Cham S, Evans MA, Denenberg JO, Golomb BA. Statin-associated muscle-related adverse effects: a case series of 354 patients. Pharmacotherapy. 2010 Jun;30(6):541-53. doi: 10.1592/phco.30.6.541. PMID 20500044
- [Background] Rallidis LS, Fountoulaki K, Anastasiou-Nana M. Managing the underestimated risk of statin-associated myopathy. Int J Cardiol. 2012 Sep 6;159(3):169-76. doi: 10.1016/j.ijcard.2011.07.048. Epub 2011 Aug 2. PMID 21813193
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Ference BA, Majeed F, Penumetcha R, Flack JM, Brook RD. Effect of naturally random allocation to lower low-density lipoprotein cholesterol on the risk of coronary heart disease mediated by polymorphisms in NPC1L1, HMGCR, or both: a 2 x 2 factorial Mendelian randomization study. J Am Coll Cardiol. 2015 Apr 21;65(15):1552-61. doi: 10.1016/j.jacc.2015.02.020. Epub 2015 Mar 11. PMID 25770315
- [Background] Ference BA, Cannon CP, Landmesser U, Luscher TF, Catapano AL, Ray KK. Reduction of low density lipoprotein-cholesterol and cardiovascular events with proprotein convertase subtilisin-kexin type 9 (PCSK9) inhibitors and statins: an analysis of FOURIER, SPIRE, and the Cholesterol Treatment Trialists Collaboration. Eur Heart J. 2018 Jul 14;39(27):2540-2545. doi: 10.1093/eurheartj/ehx450. No abstract available. PMID 29020411
- [Background] Morrone D, Weintraub WS, Toth PP, Hanson ME, Lowe RS, Lin J, Shah AK, Tershakovec AM. Lipid-altering efficacy of ezetimibe plus statin and statin monotherapy and identification of factors associated with treatment response: a pooled analysis of over 21,000 subjects from 27 clinical trials. Atherosclerosis. 2012 Aug;223(2):251-61. doi: 10.1016/j.atherosclerosis.2012.02.016. Epub 2012 Feb 16. PMID 22410123
- [Background] Yang YJ, Lee SH, Kim BS, Cho YK, Cho HJ, Cho KI, Kim SY, Ryu JK, Cho JM, Park JI, Park JS, Park CG, Chun WJ, Kim MA, Jin DK, Lee N, Kim BJ, Koh KK, Suh J, Lee SH, Lee BK, Oh SJ, Jin HY, Ahn Y, Lee SG, Bae JH, Park WJ, Lee SC, Lee HC, Lee J, Park C, Lee B, Jang Y. Combination Therapy of Rosuvastatin and Ezetimibe in Patients with High Cardiovascular Risk. Clin Ther. 2017 Jan;39(1):107-117. doi: 10.1016/j.clinthera.2016.11.014. Epub 2016 Dec 19. PMID 28007331
- [Background] Newman CB, Preiss D, Tobert JA, Jacobson TA, Page RL 2nd, Goldstein LB, Chin C, Tannock LR, Miller M, Raghuveer G, Duell PB, Brinton EA, Pollak A, Braun LT, Welty FK; American Heart Association Clinical Lipidology, Lipoprotein, Metabolism and Thrombosis Committee, a Joint Committee of the Council on Atherosclerosis, Thrombosis and Vascular Biology and Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Statin Safety and Associated Adverse Events: A Scientific Statement From the American Heart Association. Arterioscler Thromb Vasc Biol. 2019 Feb;39(2):e38-e81. doi: 10.1161/ATV.0000000000000073. PMID 30580575
- [Background] Rosenson RS, Miller K, Bayliss M, Sanchez RJ, Baccara-Dinet MT, Chibedi-De-Roche D, Taylor B, Khan I, Manvelian G, White M, Jacobson TA. The Statin-Associated Muscle Symptom Clinical Index (SAMS-CI): Revision for Clinical Use, Content Validation, and Inter-rater Reliability. Cardiovasc Drugs Ther. 2017 Apr;31(2):179-186. doi: 10.1007/s10557-017-6723-4. PMID 28421332
- [Background] Parker BA, Capizzi JA, Grimaldi AS, Clarkson PM, Cole SM, Keadle J, Chipkin S, Pescatello LS, Simpson K, White CM, Thompson PD. Effect of statins on skeletal muscle function. Circulation. 2013 Jan 1;127(1):96-103. doi: 10.1161/CIRCULATIONAHA.112.136101. Epub 2012 Nov 26. PMID 23183941
- [Background] Nissen SE, Stroes E, Dent-Acosta RE, Rosenson RS, Lehman SJ, Sattar N, Preiss D, Bruckert E, Ceska R, Lepor N, Ballantyne CM, Gouni-Berthold I, Elliott M, Brennan DM, Wasserman SM, Somaratne R, Scott R, Stein EA; GAUSS-3 Investigators. Efficacy and Tolerability of Evolocumab vs Ezetimibe in Patients With Muscle-Related Statin Intolerance: The GAUSS-3 Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1580-90. doi: 10.1001/jama.2016.3608. PMID 27039291
- [Background] Zhang H, Plutzky J, Skentzos S, Morrison F, Mar P, Shubina M, Turchin A. Discontinuation of statins in routine care settings: a cohort study. Ann Intern Med. 2013 Apr 2;158(7):526-34. doi: 10.7326/0003-4819-158-7-201304020-00004. PMID 23546564